CLINICAL TRIAL: NCT03396809
Title: The Use of Punctal Plugs in Reducing Iodine Related Ocular Surface Discomfort
Brief Title: Punctal Plugs and Iodine Related Discomfort
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution. There are no publications for this research & this is not Applicable Clinical Trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MOD00006043
Record Dates: First submitted 2017-12-20; First posted 2018-01-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye Syndromes
Keywords: punctal plugs; dry eye; ocular surface disease index
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Punctal Plugs

STUDY DESIGN:
Intervention Model Description: Investigators will be performing a case crossover study. First patients who consent will be asked to complete an Ocular Surface Disease Index (OSDI). Those whose score indicates a diagnosis of dry eye will eligible for the study. Three to five days after their intravitreal injection, patients will be contacted over the telephone and asked to complete the OSDI. At their next visit, one month later, a punctal plug will be inserted before their second injection. Three to five days after their second injection, they will be asked to complete the OSDI over the telephone. At their third visit they will receive an intravitreal injection and three to five days after they will be asked to complete a final OSDI. If patients are receiving bilateral intravitreal injections, and the OSDI survey indicates dry eyes bilaterally, then only one of the eyes will be randomly chosen for plug insertion. The other eye will then be used as a control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Punctal Plugs (Experimental): This arm of the study receives punctal plug intervention.
  Interventions: Device: Punctal plug

INTERVENTIONS:
Device: Punctal plug — Punctal plugs are FDA approved for the treatment of dry eye. They increase lubrication of the eye by blocking the drainage of tears into the lacrimal sac. The nose portion of the plug has a larger diameter which is designed to fit in the canaliculum in order to retain the plug in the punctum. The plugs will be used on-label, as it is FDA approved in the treatment of dry eye. The purpose of punctal plugs are to increase tear volume by preventing drainage of tears into the lacrimal sac. The plugs are removable if necessary. Investigators are not testing this device for effectiveness or safety.

SUMMARY:
Purpose: Intravitreal injection of medications has revolutionized the treatment microvascular diseases. These diseases often require regular, life-long injections. Ensuring patient comfort is important for compliance with long-term treatments. Patients receiving regular intravitreal injections often complain of progressive dry eye related discomfort. These symptoms are likely secondary to the use of povidone iodine as an antiseptic. Investigators hypothesize that punctal plugs could reverse the progressive ocular surface discomfort induced by povidone iodine during the post-procedural state.

DETAILED DESCRIPTION:
Retina specialists treat many diseases of the posterior segment of the eye by the delivery of medications via intravitreal injections. Many of these medications are monoclonal antibodies that need to be injected monthly. Endophthalmitis is a sight threatening complication of intravitreal injections. Limiting this complication is of primary importance in any injection protocol. The gold standard antiseptic used in intravitreal injection is Povidone-iodine (PI). PI is used to clean the surrounding ocular adnexa and is used in a 5% dilution on the ocular surface.

PI has been shown to be corrosive to the cornea, delay healing, and cause patients significant discomfort post injection especially for those with dry eye. Non-steroidal anti-inflammatories, topical anesthetics, and anticholinergics have been shown to decrease post injection discomfort1, but these measures are expensive, do not protect against corneal irritation and do not improve the healing capacity of the eye. There is a need for a cost effective measure that can reduce corneal irritation and improve healing due to the effects of PI. Punctal plugs are FDA approved for the treatment of dry eye. They increase lubrication of the eye by blocking the drainage of tears into the lacrimal sac. Our study would like to investigate the efficacy of punctal plug insertion in the prevention of dry eye symptoms caused by PI following intravitreal injection.

It has been shown that PI is toxic to the cornea at increasing concentrations. Once in contact with corneal epithelium it releases free iodine radicals causing cytotoxicity and apoptosis of cells. This makes it an effective antiseptic for Ophthalmologic procedures, but also causes significant destruction of the healthy corneal tissue2. It has also been shown in rabbits that calf serum is protective against PI induced corneal damage by providing an additional organic substrate for the PI to bind3. It is possible that natural tears can have a similar effect.

Punctal plugs are an extremely cost effective and widely used device to increase the volume of tears on the ocular surface. They block the lacrimal puncta and canalicular system that drains into the nasolacrimal duct, thereby inhibiting drainage of the natural tears into the nasal atria. In patients with dry eye who receive intravitreal injection punctal plugs may be useful in reducing corneal irritation by increasing the volume of natural tears on the ocular surface, which provides an additional organic substrate for the PI solution to bind. This has the potential to decrease the corrosive effects of the PI on the cornea, reduce healing time, and reduce pain in patients with dry eye.

Investigators will be performing a case crossover study. First patients who consent will be asked to complete an Ocular Surface Disease Index (OSDI). Those whose score indicates a diagnosis of dry eye will eligible for the study. Three to five days after their intravitreal injection, patients will be contacted over the telephone and asked to complete the OSDI. At their next visit, one month later, a punctal plug will be inserted before their second injection. Three to five days after their second injection, they will be asked to complete the OSDI over the telephone. At their third visit they will receive an intravitreal injection and three to five days after they will be asked to complete a final OSDI. If patients are receiving bilateral intravitreal injections, and the OSDI survey indicates dry eyes bilaterally, then only one of the eyes will be randomly chosen for plug insertion. The other eye will then be used as a control. There will be no blinding.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at Eye Associates of New Mexico Retina Center or the University of New Mexico Eye Clinic
* Three consecutive monthly intravitreal injections
* Patients whose OSDI score indicate dry eye (score greater than 12)
* Greater than 18 years old
* Males and Females

Exclusion Criteria:

* previous punctal plugs
* punctal cautery
* active infection
* history of ocular infection

  1. herpes simplex virus
  2. herpes zoster virus
* previous eyelid trauma

  1. surgery
  2. graft versus host disease
  3. and thyroid eye disease
* Women whom are pregnant or may become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Reduction in OSDI scores | 1 year
  For primary endpoints, investigators expect that participants will report reduced OSDI scores after intravitreal injection after insertion of punctal plug.
  The Ocular Surface Disease Index, or OSDI, is a series of 12 questions associated with a scale that assesses dry eye disease. It has three subsections that investigate the symptoms, environmental factors, and functional limitations caused by dry eye. Each question has a 5 category Likert scale associated with it with five response options that range from "none of the time" to "all of the time." The final score is calculated by multiplying the sum of the scores by 25 and dividing by the total number of questions answered. A response between 0 and 12 represents normal, 13-22 mild, 23-32 moderate, and greater than 33 severe dry eye disease. The scores range from 0-100. The OSDI scores will be conducted by Elisabeth Sledz, in person after consent and over the telephone thereafter.

SECONDARY OUTCOMES:
OSDI scores in patients receiving bilateral injections | 1 year
  Patients receiving bilateral injections will be analyzed in a subgroup. Only one of their eyes will receive a punctal plug and the other will be used as a control. OSDI scores will be completed for both eyes.
  The Ocular Surface Disease Index, or OSDI, is a series of 12 questions associated with a scale that assesses dry eye disease. It has three subsections that investigate the symptoms, environmental factors, and functional limitations caused by dry eye. Each question has a 5 category Likert scale associated with it with five response options that range from "none of the time" to "all of the time." The final score is calculated by multiplying the sum of the scores by 25 and dividing by the total number of questions answered. A response between 0 and 12 represents normal, 13-22 mild, 23-32 moderate, and greater than 33 sever dry eye disease. The scores range from 0-100. The OSDI scores will be conducted by Elisabeth Sledz, in person after consent and over the telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Nelson, COA, ROUB, Study Director — jjnelson@eyenm.com
Locations (1):
- Eye Associates of New Mexico Retina Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Georgakopoulos CD, Tsapardoni F, Makri OE. EFFECT OF BROMFENAC ON PAIN RELATED TO INTRAVITREAL INJECTIONS: A Randomized Crossover Study. Retina. 2017 Feb;37(2):388-395. doi: 10.1097/IAE.0000000000001137. PMID 27442130
- [Result] Jiang J, Wu M, Shen T. The toxic effect of different concentrations of povidone iodine on the rabbit's cornea. Cutan Ocul Toxicol. 2009;28(3):119-24. doi: 10.1080/15569520903080511. PMID 19694608
- [Result] Naor J, Savion N, Blumenthal M, Assia EI. Corneal endothelial cytotoxicity of diluted povidone--iodine. J Cataract Refract Surg. 2001 Jun;27(6):941-7. doi: 10.1016/s0886-3350(00)00750-1. PMID 11408145
- [Result] Haddock LJ, Ramsey DJ, Young LH. Complications of subspecialty ophthalmic care: endophthalmitis after intravitreal injections of anti-vascular endothelial growth factor medications. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):257-62. doi: 10.3109/08820538.2014.959616. PMID 25325851
- [Result] Jehangir N, Bever G, Mahmood SM, Moshirfar M. Comprehensive Review of the Literature on Existing Punctal Plugs for the Management of Dry Eye Disease. J Ophthalmol. 2016;2016:9312340. doi: 10.1155/2016/9312340. Epub 2016 Mar 7. PMID 27088009